CLINICAL TRIAL: NCT07293182
Title: Effect of Legs Exercises and Compression Stockings in the Prevention of Muscle Cramps Among Hemodialysis Patients
Brief Title: Legs Exercises and Compression Stockings for Prevention of Hemodialysis Muscle Cramps
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karbala University (Other)
Responsible Party: Principal Investigator, Zahraa Adel Kareem, Master's graduate student, Karbala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UOK.CON.25.091
Record Dates: First submitted 2025-12-06; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Muscle Cramp
MeSH Terms: conditions — Muscle Cramp | interventions — Stockings, Compression

STUDY DESIGN:
Intervention Model Description: participants in the Legs Exercises Group were trained to use a mini stationary bike in a supine position for 30 minute from the end of the second hour to the beginning of the third hour of hemodialysis session once per session and the same was repeated for 3 such session . The exercise was performed under the supervision of a trained nurse.
  Participants in the Compression Stockings Group: apply Compression stockings for 30 minutes from the end of the second hour to the beginning of the third hour of hemodialysis session once per session and the same was repeated for 3 such session , participants in the control group receive standard hemodialysis without legs exercises and compression stockings modalities.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- legs exercises group (Active Comparator): participants in the Legs Exercises Group were trained to use a mini stationary bike in a supine position for 30 minute from the end of the second hour to the beginning of the third hour of hemodialysis session once per session and the same was repeated for 3 such session . The exercise was performed under the supervision of a trained nurse.
  Interventions: Device: legs exercises
- compression stockings group (Active Comparator): Participants in the Compression Stockings Group: apply Compression stockings for 30 minutes from the end of the second hour to the beginning of the third hour of hemodialysis session once per session and the same was repeated for 3 such session .
  Interventions: Device: compression stockings
- control group (No Intervention): participants in the control group receive standard hemodialysis without legs exercises and compression stockings modalities.

INTERVENTIONS:
Device: legs exercises — participants in the Legs Exercises Group were trained to use a mini stationary bike in a supine position for 30 minute from the end of the second hour to the beginning of the third hour of hemodialysis session once per session and the same was repeated for 3 such session . The exercise was performed under the supervision of a trained nurse.
  Arms: legs exercises group
Device: compression stockings — Participants in the Compression Stockings Group: apply Compression stockings for 30 minutes from the end of the second hour to the beginning of the third hour of hemodialysis session once per session and the same was repeated for 3 such session .
  Arms: compression stockings group

SUMMARY:
the Objectives of this clinical trial is :

1. Investigate the effect of legs exercises in the prevention of muscle cramps among hemodialysis patients.
2. Examine the effect of compression stockings in the prevention of muscle cramps among hemodialysis patients.
3. Compare between effect of legs exercises and compression stockings in the prevention of muscle cramps among hemodialysis patients.
4. Find out the relationship between the effect of legs exercises and compression stockings in the prevention of muscle cramps with patients' demographic and clinical data.

DETAILED DESCRIPTION:
In 2023, Iraq recorded an end-stage renal disease prevalence rate of 235.6 per million, reflecting a significant increase from 2011 to 2023 . Hemodialysis (HD) is the most widely used treatment for patients with end-stage renal disease worldwide, accounting for approximately 89% of all dialysis treatments. However, HD is associated with various side effects that stem from both the dialysis procedure and the progression of the underlying disease. Among these, patients often experience muscle cramps, which manifest as severe, painful contractions affecting either a single muscle or a group of muscles . Factors triggering these cramps include electrolyte imbalances, ischemia, carnitine depletion, tissue hypoxia, hyponatremia, hypomagnesemia, fluctuations in plasma concentration, and elevated serum leptin levels . Muscle cramps negatively impact sleep and the quality of life for patients; in extreme cases, they may lead patients to consider discontinuing dialysis treatment . Additionally, shortened dialysis sessions can increase hospital admissions and the risk of mortality among dialysis patients by 13% to 30% .

Most methods for relieving muscle cramp pain have been pharmacological; however, these often elevate the risk of drug toxicity since the kidneys primarily excrete the metabolites of these drugs. This study investigates the effects of leg exercises and compression stockings on the prevention of leg cramps. These intervention methods have been less commonly utilized and have predominantly been explored in small patient populations. this research will provide insights into the effectiveness of these approaches and contribute to the development of improved prevention strategies.

When a dialysis patient exercises, the leg muscles signal the brain to increase blood flow to provide the necessary energy for activity . Exercise during dialysis positively impacts urea clearance by enhancing tissue exposure and opening blood vessels in the working muscles, allowing fluids within the tissues to flow into the intravascular space. Furthermore, ions such as potassium and phosphate move from the intracellular space into the muscle interstitial fluid during exercise, improving blood flow to the muscles and alleviating pain in these patients .

The use of graduated compression stockings applies a pressure gradient that ensures blood flows upward toward the heart rather than backing up toward the feet or sideways into the superficial veins. This application of an appropriate pressure gradient reduces the diameter of major veins, increasing the velocity and volume of blood flow. Gradient compression can effectively reverse elevated venous blood pressure, enhance skeletal muscle pumping, facilitate venous return, and improve lymphatic drainage.

ELIGIBILITY:
Inclusion Criteria:

* Those who are at least eighteen years old.
* Both genders (male & female).
* Undergoing regular hemodialysis.
* Patients who are conscious and cooperative.
* Patients experiencing muscle cramps during hemodialysis session.
* Patients who would like to participate in part in the study .
* Patients with verbally communicated skills.

Exclusion Criteria:

* Irregular hemodialysis treatment
* Presence of femoral catheters
* Any lower limb pathology or musculoskeletal impairments
* Patients undergoing emergency or first-time hemodialysis
* Pilot study participants.
* Patients decline to take part in the trial.
* Patients who are unable to tolerate the exercises and compression stockings .

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Cramp Questionnaire Chart | The intensity of muscular cramps was recorded before the hemodialysis session began and immediately at the end of the hemodialysis session.
  The instrument was developed by Morris (2014) to assess muscle cramps level. permission was obtained from the author It was translated into Arabic version by an two English-Arabic language specialist. It was used in the study to assess patients' muscle cramps level pre and post exercises and compression stockings application. This scale is composed of five features of muscle cramps: frequency, duration, pain level, leg temperature and discomfort. which was comprehensively scored as a level of muscle cramps ranging from (0-13).
Visual analogue scale (VAS) for pain | The Visual analogue scale (VAS) for pain was recorded before the hemodialysis session began and immediately at the end of the hemodialysis session.
  The Visual Analogue Scale (VAS) is a validated, subjective scale for acute and chronic pain. It was initially introduced by Hayes and Patterson in 1921. Scoring involved self-reported symptom scales that are scored with a single handwritten mark placed at a single point along a 10 cm line representing continuity between the two ends of the scale - "no pain" at the left end (0 cm) of the scale and "worst pain" at the right end of the scale (10 cm).

CONTACTS AND LOCATIONS:
Overall Officials: zahraa A Kareem, MGS, Principal Investigator — kerbala heath department

IPD SHARING:
Plan to Share IPD: No